CLINICAL TRIAL: NCT07138274
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Metyrapone in Subjects Diagnosed With Mild Autonomous Cortisol Secretion (MACS)
Brief Title: Metyrapone Study for Patients Diagnosed With Mild Autonomous Cortisol Secretion - MACS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Irina Bancos, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-007821
Record Dates: First submitted 2025-07-24; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Mild Autonomous Cortisol Secretion (MACS); Autonomous Cortisol Secretion (ACS)
Keywords: Hypercortisolism; Cortisol excess; Cushing Syndrome; Adrenal adenoma; Adrenal hyperplasia
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic; Adrenal Hyperplasia, Congenital | interventions — Metyrapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metyrapone (Experimental): Subjects in the Metyrapone arm will receive the study drug
  Interventions: Drug: Metyrapone 250 mg Oral Tablets
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive a placebo in lieu of study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metyrapone 250 mg Oral Tablets — Subjects will receive metyrapone beginning at 500 mg and titrating up to 1000 mg
  Arms: Metyrapone
Drug: Placebo — Subjects will receive placebo at 500 mg dose and titrated up to 1000 mg to match interventional arm and prevent unblinding
  Arms: Placebo

SUMMARY:
single-center, randomized, double-blind, placebo-controlled Phase 2 study to evaluate safety and efficacy of overnight metyrapone in patients with MACS.

DETAILED DESCRIPTION:
This study is a double blind, placebo-controlled phase II trial of the safety and efficacy of Metyrapone, in the treatment of MACS. Subjects will be remotely screened and interested qualified subjects will be remotely consented. Subjects will be randomized 2:1 for 6 months of the main study. At 6 months, two options will be available for subjects for months 6-12: open-label arm, observational arm.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age ≥ 18 years
4. Diagnosed with MACS i. at least 2 abnormal post-dexamethasone cortisol results1 mg post-dexamethasone cortisol >1.8 mcg/dL or ii. 8 mg post-dexamethasone cortisol >1 mcg/dL b. Historical dexamethasone suppression test results can be used if performed within 24 months prior to enrollment.
5. Adrenal imaging phenotype consistent with benign disease (adrenal adenoma/s, macronodular or micronodular adrenal hyperplasia)
6. At least one of the following comorbidities:

   1. obesity (BMI>30 kg/m2)
   2. dysglycemia
   3. dyslipidemia
   4. hypertension
   5. osteopenia
   6. osteoporosis
   7. fragility fractures
7. Ability to take oral medication and be willing to adhere to the study intervention regimen.
8. For persons of childbearing potential: : agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of ≤ 5% per year during the treatment period and for 1 month after the last dose of study treatment.
9. Stable timing for bedtime for at least one week prior to on-site study visits.
10. History of difficulty providing blood via standard blood draw methods

Exclusion Criteria:

1. Planned alternative therapy for MACS within 12 months after joining the study.
2. Current use of oral exogenous glucocorticoid therapy
3. Current use of opioid therapy >20 MME/day
4. Planned use of oral exogenous glucocorticoid therapy
5. Planned use of opioid therapy >20 MME/day
6. Use of injectable glucocorticoid within 6 weeks prior to Day 1
7. Investigator's judgement based on history/physical examination that a comorbidity or concomitant medication may impact the hypothalamic-pituitary-adrenal axis or steroid metabolome
8. Uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection
   * Symptomatic congestive heart failure
   * Unstable angina pectoris
   * Cardiac arrhythmia
   * Psychiatric illness/social situations that would limit compliance with study requirements
9. Pregnancy or lactation
10. Known allergic reactions to metyrapone
11. Suspected false positive post-dexamethasone cortisol results due to increased metabolism, poor absorption, or noncompliance with dexamethasone
12. Treatment with another investigational drug or other intervention within lower than specific therapy washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Glucocorticoid to androgen ratio | 3 and 6 months
  Glucocorticoid to androgen ratio will be calculated based on total glucocorticoids and total androgens measured through 25-steroid urine profiling.
Delta salivary cortisone | 3 and 6 months
  Waking salivary cortisone and bedtime salivary cortisone will be assessed, and delta calculated.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 0-6 months
  The investigators will assess adverse events using CTCAE v4.0 at baseline and continuously.
Change in body mass index (BMI) | 3 and 6 months
  The investigators will assess for change in the body mass index with metyrapone therapy.
Adrenal insufficiency symptoms as assessed by the AddiQoL Survey | Baseline, 1 week post dose titration, 3 and 6 months
  The investigators will administer AddiQoL Survey at baseline, 1 week after each dose titration, and at 3 and 6 months.
Adrenal insufficiency as assessed through morning ACTH and cortisol measurements. | baseline, 3, 6 months
  The investigators will measure ACTH and cortisol in the morning at baseline, 3 and 6 months to assess for biochemical adrenal insufficiency.
Improvement in hyperglycemia | 3 and 6 months
  The investigators will assess for improvement in hyperglycemia by using a composite assessment defined as: 1) decrease in fasting glucose of Hb1C, or 2) Stable biochemical measurements with a decrease in intensity of hyperglycemia therapy
Improvement in hypertension | 3 and 6 months
  The investigators will assess for improvement in hypertension using a composite assessment: 1) improvement in blood pressure measurements while on stable therapy, or 2) stable blood pressure measurements while on a lower intensity hypertension therapy.
Quality of life as assessed by SF36 form | 3 and 6 months
  The investigators will assess quality of life using SF36 at baseline, 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Bancos, MD, MS, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Yes